CLINICAL TRIAL: NCT03869229
Title: Effectiveness of Adipose-derived Mesenchymal Stem Cells in Patients With Osteoarthritis of the Knee, Hip or Glenohumeral Joint and Analysis of the Regeneration Processes Based on Inflammatory Markers, microRNAs and Clinical Features.
Brief Title: Adipose-derived Mesenchymal Stem Cells in Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002/LIFE/2019
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis; Glenohumeral Osteoarthritis; Osteoarthritis
Keywords: osteoarthritis; Adipose-derived Mesenchymal Stem Cells
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- osteoarthritis of the knee (Active Comparator): Intervention: Intra-articular injection of Adipose-derived Mesenchymal Stem Cells (ADMSC)
  Interventions: Biological: Intra-articular injection of ADMSC
- osteoarthritis of the hip (Active Comparator): Intervention: Intra-articular injection of Adipose-derived Mesenchymal Stem Cells (ADMSC)
  Interventions: Biological: Intra-articular injection of ADMSC
- osteoarthritis of the glenohumeral joint (Active Comparator): Intervention: Intra-articular injection of Adipose-derived Mesenchymal Stem Cells (ADMSC)
  Interventions: Biological: Intra-articular injection of ADMSC

INTERVENTIONS:
Biological: Intra-articular injection of ADMSC — Intervention: Intra-articular injection of Adipose-derived Mesenchymal Stem Cells (ADMSC)- ultrasound guided intra-articular injection of at least 10 million of ADMCS per procedure, maximum four procedures (i.e. injections per joint), minimum number of cells pre protocol 40 million

SUMMARY:
This phase I/II study will enroll 100 subjects with mild to moderate osteoarthritis of the hip/knee/glenohumeral joints will be enrolled according to strict inclusion and exclusion criteria. Subjects will receive a single dose of at least 10 million of autologous Adipose-derived Mesenchymal Stem Cells (ADMCS) every three months for 12 months (maximum four doses in total and at least 40 million of ADMCS in total) via ultrasound guided intra-articular injection.

DETAILED DESCRIPTION:
This phase I/II study will enroll 100 subjects with mild to moderate osteoarthritis of the hip/knee/ glenohumeral joint will be enrolled according to strict inclusion and exclusion criteria. All patients will be selected and sign consent forms, then divided into 3 groups based on clinical presentation. Participants will be exposed to abdominal liposuction procedure under local anesthesia for adipose-derived mesenchymal stem cells (ADMSC) harvesting. Stem cells will be separated from fat cells in the adipose tissue then activated in the Polish Stem Cell Bank. The activated stem cells will be injected into the knee joint via 22G spinal needle. The intra-articular stem cells injections will be performed under ultrasound guidance at the theater under spinal anesthesia. Each patient will receive a single dose of at least 10 million of ADMSC in 3 mL of normal saline every three months for 12 months (maximum four doses in total and at least 40 million of ADMSC in total) via ultrasound guided intra-articular injection. During the study period and 24 months after last injection they will be followed by clinical assessment, laboratory investigations as well as magnetic resonance imaging (MRI) of the injected joint. The local and systemic safety of the procedure and therapy with ADMSC will be also determined during study.

ELIGIBILITY:
Inclusion Criteria:

* presence of osteoarthritis of the knee, hip or glenohumeral joint
* confirmation cartilage injury, articular cartilage part or full-thickness injury by MR (Magnetic Resonance)
* joint pain of VAS (visual analog scale score) is 1 or higher while resting, 2 and higher during any physical activity
* loss of joint function based on scale specific for certain joints; for hip: HHS scale (Harris Hip Score), HOOS scale (Hip disability and Osteoarthritis Outcome Score), The Western Ontario and McMaster Universities Arthritis Index (WOMAC); for knee: modified HHS score (Harris Hip Score), The Western Ontario and McMaster Universities Arthritis Index (WOMAC), The International Knee Documentation Committee (IKDC Questionnaire) and KOOS scale (Osteoarthritis Outcome Score); glenohumeral joint: Disability of Arm, Shoulder and Hand [DASH], CONSTANT score
* clinical indication for surgical intervention
* no effect of pharmacotherapy according to The World Health Organization (WHO) analgesic ladder lasting at least 6 months
* no effect of physical rehabilitation lasting at least 6 months
* willing to participate understand and sign the consent form of this study

Exclusion Criteria:

* active inflammatory disease or infection,
* skin disease/infection around joint,
* severe heart failure,
* anemia,
* active/history of human immunodeficiency viruses (HIV), the hepatitis B virus (HBV) or the hepatitis C virus (HCV) infection,
* pregnant or breast-feeding women,
* mental disease, addiction to drugs or alcohol,
* participate other clinical experiments in 6 months,
* refuse to sign the consent form, or cannot keep follow-up visit.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-05 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
HIP DISABILITY AND OSTEOARTHRITIS OUTCOME SCORE (HOOS) | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in hip disability and osteoarthritis outcome score (HOOS) score. HOOS consists of 5 subscales: pain, other symptoms, function in activities of daily living (ADL), and function in sport and recreation (Sport/Rec), and hip-related quality of life (QOL). In total, 40 items: 10 items for pain, 5 items for other symptoms (3 for symptoms and 2 for stiff- ness), 17 items for function in ADL, 4 items for function in Sport/Rec, and 4 items for hip-related QOL. Standardized answer options are given (5 Likert boxes) and each question is scored from 0 to 4. Scores are summarized for each subscale and trans- formed to a 0-100 scale (0 indicating extreme problems and 100 indicating no problems).
Harris Hip Score | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in Harris Hip Score (HHS) score. The domains covered are pain, function, absence of deformity, and range of motion. The pain domain measures pain severity and its effect on activities and need for pain medication. The function domain consists of daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction. There are 10 items. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
Knee injury and Osteoarthritis Outcome Score (KOOS) | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in Knee injury and Osteoarthritis Outcome Score (KOOS). It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL)
  The five patient-relevant subscales of KOOS are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic assessment scales and generic measures.
modified Harris Hip Score for knee | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in modified Harris Hip Score (mHHS) score. The domains covered are pain, function, absence of deformity, and range of motion. The pain domain measures pain severity and its effect on activities and need for pain medication. The function domain consists of daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction. There are 10 items. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
The International Knee Documentation Committee (IKDC Questionnaire) | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in IKDC Questionnaire score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function
  The transformed score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
WOMAC (for hip and knee) | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in WOMAC score. WOMAC score is used to assess patients with osteoarthritis of the hip or knee using 24 parameters in 5 categories.
  1 Pain 2.Stiffness 3.Physical function 4.Social function 5. Emotional function
  Scoring and Interpretation
  Response : points none - 0 slight 1 moderate 2 severe 3 extreme 4
  score = = summary (points for relevant items) average score = = (total score) / (number of items) Interpretation: minimum total score: 0 maximum total score: 96 minimum pain subscore: 0 maximum pain subscore: 20 minimum stiffness subscore: 0 maximum stiffness subscore: 8 minimum physical function subscore: 0 maximum physical function subscore: 6
Disability of Arm, Shoulder and Hand [DASH] | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in DASH score. DASH outcome measure is a 30-item. The items enquire about the degree of difficulty in performing different physical activities because of arm, shoulder and hand problems (21 items), the severity of each of the symptoms of pain, activity-related pain, tingling, weakness and stiffness (five items) and the impact of the problem on social functioning, work, sleep and self-image (four items).
  The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability
  A minimum score is 30; a maximum is 150. The range of the scores, therefore-from 30 to 150-equals 120. The raw score is then transformed to a zero-to-100 scale with zero reflecting no disability (good function) and 100 reflecting maximum disability.
The Constant-Murley score (CMS) | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in CMS score. CMS is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient
  The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
Visual Analog Scale (VAS) | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Change in Visual Analog Scale (VAS) for pain in the target hip following completion of treatment cycles. Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control The VAS is a commonly used tool in health outcome studies, when using it to assess importance of certain action or intervention, how we can interpret the results, on 1 to 10 line (where 1; the least and the 10; the highest)

SECONDARY OUTCOMES:
Nature, incidence and severity of adverse events (AEs) | Time Frame: Baseline (T0), 3 months (T1), 6 months (T2), 9 months (T3), 12 months (T4), 24 months (T5)
  Defined as any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline (i.e., if present upon study entry) during the study regardless of causal relationship.
  Methods i. Spontaneous subject reports ii. Subject interview by study personnel iii. Clinical examination during face-to-face clinic follow-ups. Defined as any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline (i.e., if present upon study entry) during the study regardless of causal relationship.
  Methods i. Spontaneous subject reports ii. Subject interview by study personnel iii. Clinical examination during face-to-face clinic follow-ups
Change in cartilage thickness | Baseline, and 12 months post-treatment cycle
  Cartilage thickness on MRI in mm
Change in cartilage volume | Baseline, and 12 months post-treatment cycle
  Cartilage volume on MRI in ml
Change in cartilage morphology | Baseline, and 12 months post-treatment cycle
  Cartilage morphology on MRI. Change in the International Cartilage Repair Society (ICRS) classification. It is based on grading of cartilage lesions, in which lesions are graded 0 to 4 based on depth of the lesion. Grade 1 and 2 lesions have excellent prognosis. Grade 2 and 3 lesions may benefit from cartilage debridement or other more conservative surgical measures. Grade 4 lesions extend into the subchondral bone and may require bone grafting if bony cavitation is extensive
Change in subchondral bone morphology | Baseline, and 12 months post-treatment cycle
  Subchondral bone morphology (i.e. edema) on MRI
Inflammation monitoring | Baseline, and 12 months post-treatment cycle]
  Baseline, and 12 months post-treatment cycle based on changes of concentrations of interleukin (IL)-1β (pg/ml), IL-6 (pg/ml), IL-8 (pg/ml), IL-11 (pg/ml), tumor necrosis factor (TNF)-alpha (pg/ml)
Inflammation monitoring | Baseline, and 12 months post-treatment cycle
  Baseline, and 12 months post-treatment cycle based on changes of concentrations of CD40L (ng/ml)
Inflammation monitoring | Baseline, and 12 months post-treatment cycle
  Baseline, and 12 months post-treatment cycle based on changes of high-sensitivity C-reactive protein (hsCRP ) (mg/dl)
Inflammation monitoring | Baseline, and 12 months post-treatment cycle
  Baseline, and 12 months post-treatment cycle based on changes of miRNA expression (ug/dl) defined on microarray profiling

CONTACTS AND LOCATIONS:
Overall Officials: Marek Postula, MD, PhD, Principal Investigator — Medical University of Warsaw; Robert Smiegielski, MD, Study Director — Life Clinic
Locations (1):
- Life Clinic, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: No